CLINICAL TRIAL: NCT06278350
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of D-2570 in Participants With Moderate-to-Severe Plaque Psoriasis
Brief Title: Evaluate the Efficacy and Safety of D-2570 in Participants With Moderate-to-Severe Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: InventisBio Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D2570-201
Record Dates: First submitted 2024-01-30; First posted 2024-02-26 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- D-2570 group 1 (Experimental): D-2570 group 1
  Interventions: Drug: D-2570
- D-2570 group 2 (Experimental): D-2570 group 2
  Interventions: Drug: D-2570
- D-2570 group 3 (Experimental): D-2570 group 3
  Interventions: Drug: D-2570
- Placebo group (Placebo Comparator): Placebo group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: D-2570 — Randomized in a 1:1:1:1 ratio through the randomization system, and assigned to D-2570 group
  1, group 2, group 3 or placebo group.
  Arms: D-2570 group 1; D-2570 group 2; D-2570 group 3
Drug: Placebo — Randomized in a 1:1:1:1 ratio through the randomization system, and assigned to D-2570 group
  1, group 2, group 3 or placebo group.
  Arms: Placebo group

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multicenter clinical trial in participants with moderate-to-severe plaque psoriasis .

ELIGIBILITY:
Inclusion Criteria:

1. Subject voluntarily takes part in the study after being fully informed,signs a written ICF, and agrees to follow procedures specified in the study protocol;
2. Plaque psoriasis assessed by the investigator as suitable for systemic treatment and stable (defined as stable as no significant outbreak of morphological change or disease activity assessed by the investigator) for at least 6 months prior to signing informed consent;
3. During the screening period and before taking the investigational drug for the first time, psoriatic surface area (BSA) ≥10%, PGA score ≥ 3, PASI score ≥ 12;
4. Hematology, Blood chemistry and Urinalysis examination were basically normal.

Exclusion Criteria:

1. Erythrodermic psoriasis, pustular psoriasis, guttate psoriasis, reverse psoriasis, drug-induced psoriasis;
2. Have other skin lesions that affect the evaluation of treatment outcomes, such as eczema;
3. History of herpes zoster/herpes simplex, or presence of herpes zoster/herpes simplex infection during the screening period;
4. Have a history of tuberculosis, or active tuberculosis, or latent tuberculosis, or suspected clinical manifestations of tuberculosis infection;
5. Other conditions that the investigator considers inappropriate for participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with at least 75% improvement in PASI | Day 1-Day 85
  Percentage of subjects with at least 75% improvement in PASI from baseline at week 12 of treatment

SECONDARY OUTCOMES:
Percentage of subjects with at least 75% improvement in PASI | Day 1-Day 56
  Percentage of subjects with at least 75% improvement in PASI from baseline at weeks 4 and 8 of treatment;
Percentage of subjects with at least 90% improvement in PASI | Day 1-Day 85
  Percentage of subjects with at least 90% improvement in PASI from baseline at weeks 4, 8, and 12 of treatment;
Percentage of subjects with 100% improvement in PASI | Day 1-Day 85
  Percentage of subjects with 100% improvement in PASI from baseline at weeks 4, 8, and 12 of treatment;
Percentage improvement in PASI | Day 1-Day 85
  Percentage improvement in PASI from baseline at weeks 4, 8, and 12 of treatment;
Percentage of subjects with a PGA | Day 1-Day 85
  Percentage of subjects with a PGA score of 0 or 1 at weeks 4, 8, and 12 of treatment;
The main PK parameters ：Time to maximum measured plasma concentration（Tmax） | Day 1-Day 85
  The main PK parameters ：Time to maximum measured plasma concentration（Tmax）
The main PK parameters ：Peak Plasma Concentration（Cmax) | Day 1-Day 85
  The main PK parameters ：Peak Plasma Concentration（Cmax）
The main PK parameters：Area under the plasma concentration versus time curve（AUC） | Day 1-Day 85
  The main PK parameters：Area under the plasma concentration versus time curve（AUC）
The main PK parameters：Vz/F (apparent volume of distribution) | Day 1-Day 85
  The main PK parameters：Vz/F (apparent volume of distribution)
The main PK parameters： Half-life（t1/2） | Day 1-Day 85
  The main PK parameters： Half-life（t1/2）
The main PK parameters： Mean Residence Time (MRT) | Day 1-Day 85
  The main PK parameters： Mean Residence Time (MRT)
The main PK parameters：CL/F (apparent clearance) | Day 1-Day 85
  The main PK parameters：CL/F (apparent clearance)
Weight and height will be combined to report BMI in kg/m^2 | Day -28-Day 99
  Weight and height will be combined to report BMI in kg/m^2
Incidence and severity of AEs based on NCI CTCAE V5.0 | Day -28-Day 99
  Incidence and severity of AEs based on NCI CTCAE V5.0
Incidence and severity of TEAEs based on NCI CTCAE V5.0 | Day -28-Day 99
  Incidence and severity of TEAEs based on NCI CTCAE V5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhong Zhang, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No